CLINICAL TRIAL: NCT00255372
Title: Polyethylene Glycol Laxative (Macrogol 4000;Forlax®) for Treatment of Chronic Constipation in Children : A Phase III, Bicentric, Randomized, Double-blind, Lactulose Controlled Study.
Brief Title: To Determine the Effect of Forlax® Treatment in Children With Chronic Constipation Who May Also Suffer From Soiling/ Faecal Incontinence.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-38-52072-012
Record Dates: First submitted 2005-11-17; First posted 2005-11-18 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Chronic Constipation
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: PEG 4000 (Forlax®)
- 2 (Active Comparator)
  Interventions: Drug: Lactulose active and Lactulose placebo

INTERVENTIONS:
Drug: PEG 4000 (Forlax®) — Powder for oral solution. 2 sachets of 4g, from baseline every two weeks over a 4 week treatment period.
  Arms: 1
Drug: Lactulose active and Lactulose placebo — Powder for oral solution. 1 sachet of 3.3g lactulose active and 1 sachet of lactulose placebo. From baseline every two weeks over a 4 week treatment period.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Forlax® is more effective than placebo in relieving chronic constipation in children who may also suffer from soiling or faecal incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Chronic constipation (defined as at least 3 months of less than 2 bowel movements (BMs) per week and/or one of the following symptoms : hard stool, painful defecation, encopresis)
* Constipation previously treated by dietary advice (high fiber diet) for at least two weeks without efficacy

Exclusion Criteria:

* Organic bowel diseases
* Suspected GI obstruction
* History of GI surgery

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2005-04; Primary Completion 2008-05-20 (Actual); Study Completion 2008-05-20 (Actual)

PRIMARY OUTCOMES:
Bowel movement frequency | week 4

SECONDARY OUTCOMES:
Subjective symptoms associated with defecation. | At every visit

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (2):
- Thailand (2):
  - Ramathibodi Hospital, Mahidol University,, Bangkok
  - Maharat Nakhon Ratchasima Hospital, Nakhon Ratchasima

REFERENCES:
- [Derived] Treepongkaruna S, Simakachorn N, Pienvichit P, Varavithya W, Tongpenyai Y, Garnier P, Mathiex-Fortunet H. A randomised, double-blind study of polyethylene glycol 4000 and lactulose in the treatment of constipation in children. BMC Pediatr. 2014 Jun 19;14:153. doi: 10.1186/1471-2431-14-153. PMID 24943105